CLINICAL TRIAL: NCT04563884
Title: Validity of the French Version of Deafness Questionnaires for Children and Adolescents
Acronym: SSQ-PEACH
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200794; 2020-A01274-35 (Other: ID RCB number)
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Deafness
Keywords: Deafness; Children; SSQ questionnaire; PEACH questionnaire
MeSH Terms: conditions — Deafness | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with deafness: Patients aged 12 months to 17 years with deafness
  Interventions: Other: Questionnaires
- Controls: Normal-hearing patients aged 12 months to 17 years
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Children 12 months to 5 years old will receive PEACH alone, children 5 years old to 11 years old will receive PEACH and SSQ-P, and children and adolescents over 11 years old will receive SSQ-P and SSQ-C (even between 11 and 13 years old, the PEACH also).
  Questionnaires will be completed twice, 15 days apart.
  Other Names: The Parents' Evaluation of Aural/Oral Performance of Children (PEACH). The Speech, Spatial and Qualities of Hearing Scale (SSQ)

SUMMARY:
The care of deafness in children is difficult and the relevance of interventions is difficult to evaluate based on audiometric measurements alone.

Generic pediatric quality of life tools have been validated and used, among other things, to assess the quality of life of children with deafness. However, these non-specific tools do not make it possible to precisely target which factors and interventions are the most important for the quality of life in this population.

Achieving a score to monitor the quality of life objectively over time is fundamental to verify the effectiveness of interventions, and assess the impact on the child. There is currently no validated test in French for any of these uses and populations.

The objective of the study is to adapt the questionnaires "PEACH", "SSQ child (SSQ-C)" and "SSQ parents (SSQ-P)" to the French child, and statistically measure their internal and external validity by comparing them to a control group.

The validation of these three tests (PEACH, SSQ-P, SSQ-C) would make it possible to assess the hearing performance and quality of life of almost the entire pediatric population, for use in both clinical and academic practice.

DETAILED DESCRIPTION:
Neonatal sensorineural hearing loss is a frequent pathology, affecting around 800 newborns per year in France, or an incidence of 0.8 to 1.3 per 1000 births, comparable to other industrialized countries. It can affect the development of speech and language and lead to impaired quality of life.

Studies have shown that children with hearing loss score lower on general quality-of-life measurement tools, compared to their normal-hearing peers. A poorer quality of life in patients with sensorineural hearing loss may also reflect physical, academic, social or emotional difficulties. They are also exposed to an increased risk of poor development of language and social skills, as well as an increased risk of developing psychiatric pathologies.

The care of deafness in children is difficult and the relevance of interventions is difficult to evaluate based on audiometric measurements alone.

Generic pediatric quality of life tools have been validated and used, among other things, to assess the quality of life of children with deafness. However, these non-specific tools do not make it possible to precisely target which factors and interventions are the most important for the quality of life in this population.

Achieving a score to monitor the quality of life objectively over time is fundamental to verify the effectiveness of interventions, and assess the impact on the child. There is currently no validated test in French for any of these uses and populations.

The Parents' Evaluation of Aural/Oral Performance of Children (PEACH) is a hetero-evaluation score used to study the quality of a child's communication from an early age (from 4 months in some studies) and up to 13 years. This tool is specifically designed for children with hearing aids or a cochlear implant. It has been translated into Swedish and Spanish and used in numerous international publications.

The Speech, Spatial and Qualities of Hearing Scale (SSQ) is an adult self-assessment score assessing, in three categories, the performance of speech comprehension, spatial hearing and hearing quality. It is widely used internationally in its adult version.

This adult score has been adapted and used for the pediatric population in a hetero-evaluation score by parents (SSQ-P) from 5 years old, and a simplified score (SSQ-C) usable by children> 11 years.

In addition, the authors of the adult SSQ also prepared and validated a Handicap questionnaire to target the impact of hearing loss on quality of life, and integrated into the SSQ self-assessment.

The objective of the study is to adapt the questionnaires "PEACH", "SSQ child (SSQ-C)" and "SSQ parents (SSQ-P)" to the French child, and statistically measure their internal and external validity by comparing them to a control group.

The validation of these three tests (PEACH, SSQ-P, SSQ-C) would make it possible to assess the hearing performance and quality of life of almost the entire pediatric population, for use in both clinical and academic practice.

ELIGIBILITY:
Inclusion Criteria:

* Minors aged 12 months to 17 years (inclusive)
* Patients followed in consultation at Necker Hospital in the Pediatric ENT department
* holders of parental authority not opposed to participation in the study

Patients :

* Patients with deafness with mean tonal thresholds of at least 30dB, uni- or bilateral
* Perceptual or transmission deafness or mixed

Controls:

* Patients not presenting a hearing disorder at the time of inclusion or in his or her history
* Examination of the normal eardrums
* No history of ear surgery

Exclusion Criteria:

* Psychomotor retardation
* Abnormal neurological examination
* Mother tongue of the child and parents other than French

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients followed by the Pediatric ENT department of Necker-Enfants Malades hospital.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-10-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Paired student t-test | 1 year
  Reproducibility of the questionnaire completed by a subject at 15 days apart
Cronbach alpha test | 1 year
  Internal consistency
Item-total Pearson correlation | 1 year
  Measure of reliability
Principal components analysis | 1 year
  Measure of efficiency
Receiver Operating Characteristic (ROC) curve | 1 year
  Limit value of normality

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Denoyelle, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gargula S, Simon F, Celerier C, Couloigner V, Leboulanger N, Loundon N, Denoyelle F. French adaptation and validation of parents' evaluation of aural/oral performance of children (PEACH) scale in children. Int J Audiol. 2023 Jun;62(6):592-598. doi: 10.1080/14992027.2022.2059714. Epub 2022 May 9. PMID 35533092